CLINICAL TRIAL: NCT04756739
Title: Menstrual Cycle Symptom Tracking Study
Brief Title: Menstrual Cycle Symptom Tracking
Status: Completed | Type: Observational
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTOCOL-1276
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Menstrual Cycles

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Clearblue Connected Ovulation Test System — Clearblue Connected Ovulation Test System which is a CE marked device used for tracking the menstrual cycle

SUMMARY:
This study will provide menstrual cycle symptom information from women over the course of three menstrual cycles to determine whether there are any noticeable physiological changes that can be related to stage of the menstrual cycle or onset of menstruation.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18 years and over
* Regular menstrual cycles
* Owns a compatible smart phone i.e. iPhones® and AndroidTM phones equipped with Bluetooth® 4.0/BLE
* Willing to use their own smartphone for the duration of this study and to download and install the study app
* Willing to give informed consent

Exclusion Criteria:

* Currently trying to conceive
* Currently or recently pregnant or breastfeeding
* Taking any treatment which may affect the menstrual cycle (e.g. contraceptive pill, fertility medications or hormone replacement therapy)
* Taking or undergoing any other medical treatment for fertility such as ovulation drugs, artificial insemination and assisted fertility such as In vitro fertilization (IVF) or Intracytoplasmic sperm injection (ICSI)
* Has abnormal liver or kidney function
* Taking antibiotics containing tetracycline
* Taking clomiphene citrate or other ovulation induction drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female only
Study Population: Healthy, female volunteers
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Menstrual Cycle Symptoms | 3 months
  The primary objective of this study is to collect information from women on their experience of menstrual cycle symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Johnson, PhD, Study Director — SPD Development Company
Locations (1):
- SPD Development Company Ltd, Bedford, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD